CLINICAL TRIAL: NCT06367517
Title: Efficacy and Safety of Tocilizumab in Patients With Active Moderate-to-Severe Corticosteroid-Resistant Thyroid Eye Disease: Open, Prospective, Observational Study
Brief Title: Tocilizumab in Corticosteroid-Resistant Graves' Orbitopathy (Thyroid Eye Disease)
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Tomasz Bednarczuk, Prof, Medical University of Warsaw
Other Study IDs: KB/114/2022
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Orbitopathy, Graves; Thyroid Eye Disease; Ophthalmopathy
Keywords: Graves' disease; Graves' orbitopathy; Tocilizumab; Thyroid Eye Disease; Hyperthyroidism
MeSH Terms: conditions — Graves Ophthalmopathy; Eye Diseases; Graves Disease; Hyperthyroidism | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graves' orbitopathy: Patients with active, moderate to severe TED, without disease improvement after methylprednisolone pulse therapy in an intermediate-dose schedule (starting dose of 0.5 g once weekly for 6 weeks, followed by 0.25 g once weekly for 6 weeks) or high-dose regimens (a starting dose of 0.75 g once weekly for 6 weeks, followed by 0.5 g once weekly for 6 weeks) with or without concomitant radiotherapy.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab administrated at a dose of 8 mg/kg, given once every four weeks
  Other Names: RoActemra

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Tocilizumab as second/third line treatment in patients with Active Moderate-to-Severe Corticosteroid-Resistant Thyroid Eye Disease.

DETAILED DESCRIPTION:
Graves' Orbitopathy (GO) is an autoimmune disease that involves orbital tissues, leading to temporary or permanent damage to the eye. Although GO is a rare condition, it negatively affects the quality of life in the majority of patients. In the majority of european centers, high-dose intravenous glucocorticoid (GCs) therapy remains the first-line treatment in patients with active, moderate-to-severe GO. However, GCs are effective in only 45-60% of patients, with a high probability of diseases relapse (10-40%) or disease progression to dysthyroid optic neuropathy (up to 10%). Due to limited efficacy of GCs, unpredictable relapses and progression of GO, the management of GO remains a challenge.

A few studies have demonstrated that interleukin-6 (IL-6) blockade with tocilizumab (TCZ) is effective in GC-refractory GO. However, the long-term outcomes of TCZ remain scarce.

Therefore, the investigators are planning to assess the therapy with Tocilizumab, regarding clinical outcomes and adverse events. The investigators plan to include a total of 30 patients with active, moderate-to-severe, corticosteroid-resistant GO over a period of approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female, 18-80 years old
* Patients with active (Clinical Activity Score ≥ 3 in 7-item scale) and moderate-to-severe GO, diagnosed according to the EUGOGO guidelines, after the completion of MP pulse treatment, WITH

  o Deterioration of GO (in 1 or 2 eyes) when two of the following occurred:
* increase in palpebral aperture by at least 2 mm;
* deterioration in CAS by at least 2 points (7-point CAS)
* increase in exophthalmos by at least 2 mm;
* worsening of diplopia (appearance or change in the degree)
* worsening in ocular motility by 8o

  o Incomplete response in both eyes to intravenous methylprednisolone pulse therapy; defined changes smaller than previously defined in any of the mentioned parameters.
* Euthyroid for at least 6-8 weeks (serum free hormone concentrations within 30% of normal range) on either anti-thyroid medications (tyonamides) to control hyperthyroidism or L-thyroxine for replacement therapy for hypothyroidism.
* Negative pregnancy test in women of fertile age.
* All female patients of fertile age must use a reliable contraceptive method to prevent pregnancy during the study period, and at least during a period of six months following the last dose of the investigational medicinal product.

Exclusion Criteria:

* Signs of sight-threatening TED (severe keratopathy, optic neuropathy)
* Pregnant or breastfeeding woman or woman planning to become pregnant during the study
* Patients who could need treatment with radioactive iodine or thyroidectomy during the study
* Treatment with any biological therapy at any time.
* Active infection.
* History of recurrent clinically significant infection or recurrent bacterial infections.
* Positive quantiferon without documentation of treatment for tuberculosis (TB) infection or documentation of no need for such therapy.
* Required management of infections, as follows: currently on any suppressive therapy for a chronic infection, hospitalization for treatment of infection within 60 days before Day 0, use of parenteral antibiotics within 60 days before Day 0, use of oral antibiotics within 30 days before Day 0.
* History of intestinal ulceration or diverticulitis
* Patients with a history of chronic liver disease or liver disorders: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) above 5 times upper limit of normal (ULN)
* HBsAg positive test.
* HBcAb positive test, regardless of HBsAb status, will undergo HBV DNA which, if positive, will be excluded. HbcAb positive, HbsAg negative patients with undetectable HBV DNA will receive antiviral prophylaxis throughout the immunosuppressive therapy.
* Hepatitis C antibody positive test at screening.
* Positive test for Human Immunodeficiency Virus (HIV) antibody at screening or historically. Denied consent to HIV testing.
* Absolute neutrophil count (ANC) < 2.0 × 109/L or a platelet count < 100×103/μL
* Alkaline phosphatase and bilirubin>1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is<35%).
* Cardiovascular or cerebrovascular disease clinically significant.
* Other serious chronic illness (including uncontrolled diabetes mellitus, renal disease, pulmonary disease, major depression).
* History of sarcoidosis.
* Primary or secondary immunodeficiency.
* History of IgE-mediated or non-IgE-mediated hypersensitivity.
* History of reactions or anaphylactic allergic severe human monoclonal antibodies, humanized or murine.
* Administration of live vaccines given within 30 days prior to administration of (Day 0) or concurrently with tocilizumab (during study).
* Splenectomy.
* Current drug or alcohol abuse or dependence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with active, moderate-to-severe Graves' orbitopathy (GO), resistant to corticosteroid treatment, will be enrolled to participate in the study. They will be diagnosed and treated at a tertiarry referall center.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Disease improvement | at 16, 24 and 48 weeks
  Proportion of patients improved at 16, 24 and 48 weeks as assessed by a composite ophthalmic score. A response to treatment will be considered positive in the case of an improvement of at least 2 of the following features in 1 eye, without concomitant deterioration in the other eye:
  * decrease in eyelid aperture by at least 2 mm measured with a ruler
  * decrease in proptosis by at least 2 mm measured with Hertel Exophthalmometer
  * increase in eyelid motility by at least 8° assessed by ophthalmologist or improvement of Bahn-Gorman diplopia score (Grade I - intermittent diplopia, Grade II - Inconstant diplopia, Grade III - Constant diplopia)
  * decrease in 7-item (spontaneous retrobulbar pain, pain on attempted upward or downward gaze, redness of eyelids, redness of conjunctiva, sweeling of caruncle or plica, swelling of eyelids, swelling of conjunctiva) clinical activity score (CAS) by at least 2 points.
Improvement of quality of life | at 16, 24 and 48 weeks
  Improvement of quality of life according to the disease-specific quality of life questionnaire in Graves' orbitopathy (GO-QoL) at 16, 24 and 48 weeks. All Go-QoL questions will be scored as 'severely limited' (one point), a 'little limited' (two points), or 'not limited at all' (three points). The questions will be transformed from 0 to 100 by the following formula: total score= (raw score- 8)/16 x100. An improvement in QoL wil be considered, if there will be an increase of 6 or more points on either one (or both) the GO-QoL scales (functioning and appearance);

SECONDARY OUTCOMES:
Disease inactivation | at 16, 24 and 48 weeks
  Proportion of patients achieving response in reduction of clinical activity score (CAS) defined as reduction of ≥ 2 points from baseline in the study eye without deterioration (≥ 2 point increase) of CAS in the fellow eye
Proportion of patients achieving response in specific GO signs and symptoms | at 16, 24 and 48 weeks
  * reduction of proptosis of least 2 mm without deterioration (≥ 2 mm increase) of proptosis in the fellow eye measured with Hertel Exophthalmometer.
  * diplopia; proportion of participants with baseline diplopia > 0 and a reduction of ≥ 1 grade assessed according to Bahn-Gorman diplopia score (Grade I - intermittent diplopia, Grade II - Inconstant diplopia, Grade III - Constant diplopia)
  * ocular motility; an increase of at least 8° assessed by ophthalmologist
  * palpebral aperture; an increase of at least 2 mm measured with a ruler
  * reduction in spontaneous or gaze-evoked retrobulbar pain - a binary scale (yes/no)
  * reduction in swelling of eyelids (severe/moderate/mild), redness of eyelids (yes/no), redness of conjunctiva (yes/no), sweeling of caruncle or plica (yes/no), swelling of conjunctiva (yes/no)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | from 0 to 16 weeks
  Incidence of adverse events, with severity determined according to NCI CTCAE v5.0
Decrease in concentration of thyrotropin receptor antibodies | at 4, 8, 12, 16, 24 and 48 weeks
  Decrease in concentration of thyrotropin receptor antibodies
Decrease in levels of proinflammatory cytokines | at 4, 8, 12, 16, 24 and 48 weeks
  Decrease in serum levels of interleukin-17a and interleukin-23
Number of the rehabilitative surgeries performed after immunosuppressive therapy | at 48 weeks
  Rehabilitative surgery includes orbital decompression, squint surgery, lid lengthening, and blepharoplasty/browplasty
The rate of disease relapse | at 48 weeks
  Proportion of patients with worsening of symptoms associated with GO after a period of improvement or stability. The relapse of the disease will be noted in case of a deterioration of at least 2 of the following features in 1 eye:
  * increase in eyelid aperture by at least 2 mm measured with a ruler ,
  * increase in exophthalmos by at least 2 mm measured with Hertel Exophthalmometer,
  * decrease in eyelid motility by at least 8° assessed by ophthalmologist or deterioration of ≥ 1 grade in Bahn-Gorman diplopia score (Grade I - intermittent diplopia, Grade II - Inconstant diplopia, Grade III - Constant diplopia),
  * increase in 7-item (spontaneous retrobulbar pain, pain on attempted upward or downward gaze, redness of eyelids, redness of conjunctiva, sweeling of caruncle or plica, swelling of eyelids, swelling of conjunctiva) clinical activity score (CAS) by at least 2 points.
Decrease in proptosis by at least 2 mm assessed using magnetic resonance imaging (MRI) | at 16 weeks
  Measurement of exophthalmos (the distance between the interzygomatic line and the anterior surface of the globe - corneal apex) on axial T2W orbital MRI images performed at week 16 in comparison to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Bednarczuk, MD, PHD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine and Endocrinology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Individual data will be provided at request

REFERENCES:
- [Background] Burch HB, Perros P, Bednarczuk T, Cooper DS, Dolman PJ, Leung AM, Mombaerts I, Salvi M, Stan MN. Management of Thyroid Eye Disease: A Consensus Statement by the American Thyroid Association and the European Thyroid Association. Thyroid. 2022 Dec;32(12):1439-1470. doi: 10.1089/thy.2022.0251. Epub 2022 Dec 8. PMID 36480280
- [Background] Perez-Moreiras JV, Gomez-Reino JJ, Maneiro JR, Perez-Pampin E, Romo Lopez A, Rodriguez Alvarez FM, Castillo Laguarta JM, Del Estad Cabello A, Gessa Sorroche M, Espana Gregori E, Sales-Sanz M; Tocilizumab in Graves Orbitopathy Study Group. Efficacy of Tocilizumab in Patients With Moderate-to-Severe Corticosteroid-Resistant Graves Orbitopathy: A Randomized Clinical Trial. Am J Ophthalmol. 2018 Nov;195:181-190. doi: 10.1016/j.ajo.2018.07.038. Epub 2018 Aug 4. PMID 30081019
- [Background] Rymuza J, Kus A, Bialas-Niedziela D, Turczynska M, Kecik D, Bednarczuk T. Long-term remission of corticosteroid-resistant Graves' orbitopathy after therapy with tocilizumab. Endokrynol Pol. 2024;75(1):117-118. doi: 10.5603/ep.97224. PMID 38497401
- [Background] Bartalena L, Kahaly GJ, Baldeschi L, Dayan CM, Eckstein A, Marcocci C, Marino M, Vaidya B, Wiersinga WM; EUGOGO dagger. The 2021 European Group on Graves' orbitopathy (EUGOGO) clinical practice guidelines for the medical management of Graves' orbitopathy. Eur J Endocrinol. 2021 Aug 27;185(4):G43-G67. doi: 10.1530/EJE-21-0479. PMID 34297684
- [Background] Sawicka-Gutaj N, Bednarczuk T, Daroszewski J, Waligorska-Stachura J, Miskiewicz P, Sowinski J, Bolanowski M, Ruchala M. GO-QOL--disease-specific quality of life questionnaire in Graves' orbitopathy. Endokrynol Pol. 2015;66(4):362-6. doi: 10.5603/EP.2015.0046. PMID 26323474